CLINICAL TRIAL: NCT04477720
Title: HCC Observation Study
Brief Title: Retrospective Analysis of De-identified Deceased HCC Patients
Status: Completed | Type: Observational
Sponsor: Carr, Brian (Other)
Responsible Party: Sponsor
Other Study IDs: BCarr
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2020-07

CONDITIONS: Survival
Keywords: HCC, AFP, MTD, survival, NLR, PLR, Tumor Aggressiveness
MeSH Terms: conditions — Metatropic dwarfism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
De-identified deceased HCC patients who were not surgical candidates were evaluated for their clinical baseline characteristics associated with their survival. Baselines included tumor markers, blood counts and liver function tests and CAT-scan based tumor size and numbers and presence of portal vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven HCC

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Yes
Study Population: Patients presenting for HCC management
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 1995-06 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Survival | 10 years
  Overall survival

IPD SHARING:
Plan to Share IPD: Undecided